CLINICAL TRIAL: NCT04025255
Title: A 28-day, Randomized, Double-Blind, Placebo Controlled Study of the Nutritional Supplement Braini for Support of Brain Health in Healthy Younger and Older Adults Based on Performance on Standard Memory and Cognitive Performance Assays
Brief Title: The Memory and Cognitive Performance Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vita Naturel, LLC (Industry)
Collaborators: University of North Carolina at Asheville (Other); Braini LLC (Industry); University of South Alabama (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 1428244-1
Record Dates: First submitted 2019-07-16; First posted 2019-07-18 (Actual); Last update posted 2022-11-21 (Actual); Status verified 2022-11

CONDITIONS: Cognitive Function; Memory; Brain Health
Keywords: Brain Health; Cognitive Abilities; Mental Orientation; Short-term Memory; Executive Function
MeSH Terms: conditions — Orientation, Spatial

STUDY DESIGN:
Intervention Model Description: Randomized, double-blind, placebo-controlled study
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Participants and study personnel will be blinded to group assignment. Study personnel will receive 24 bottles each of either "active" or "placebo" product from the supplier. The bottles would be numbered sequentially from 101 to 148 for the younger cohort and 201 to 248 for the older cohort. Within that sequence, randomized blocks of 4 bottles each would be filled with either "active" or "placebo" product, for a total of 12 blocks. The bottler will not reveal to anyone which bottles got filled with which type of product until after the conclusion of the trial. Except for having a different sequential number on the label, the bottles will be indistinguishable.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Braini (Experimental): 28-day oral capsules of Braini
  Interventions: Dietary Supplement: Braini
- Placebo (Placebo Comparator): 28-day oral capsule of placebo comparator
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Braini — A novel, neuro-protective and neuro-restorative dietary supplement composed of a combination of active ingredients which have been commercially-available since at least 2015 or have achieved FDA new dietary ingredient notification (NDIN) status in 2018
  Arms: Braini
Dietary Supplement: Placebo — Matched placebo
  Arms: Placebo

SUMMARY:
The primary purpose of this study is to evaluate the impact of a novel, neuro-protective and neuro-restorative dietary supplement (Braini®) on standardized memory and cognitive performance parameters. The principal active ingredients in the Braini® supplement have been commercially-available since at least 2015 or have achieved FDA new dietary ingredient notification (NDIN) in 2018, with no adverse events reported to the FDA.

A 28-day randomized, double-blinded, placebo-controlled dietary supplement study will be conducted with a cohort of younger and a cohort of colder adults to achieve the purpose of this study. The research team hypothesizes that Braini® will improve standardized performance scores measured by CNS Vital Signs standard memory and cognitive performance assays more effectively than placebo.

DETAILED DESCRIPTION:
The number of people affected by cognitive decline continues to rise as the US population ages. A recent report indicates that this decline can be seen as early as age 45. Optimizing cognitive function during adulthood is a key mechanism to combat cognitive decline as one reaches older adulthood.

Recent advances in cognitive wellness management have shown that tailored diet and lifestyle regimens that factor in various biomarkers and proclivities signaling cognitive decline (e.g. family genetics) can cause a person with a declining MOCA (measure of cognitive ability) score to restore or achieve an improved MOCA score.

A number of clinical trials have studied nutraceutical ingredients for improved memory enhancement and/or cognitive performance. While the individual ingredients are already well-utilized in commerce globally, the Braini® formulation is novel, harnessing synergistic effects seen in a new in vitro human neural cell challenge study carried out in South Korea by the study sponsor. In this study a series of independent in vitro (cell line) tests of the active nutraceutical constituents that comprise the Braini® dietary supplement product line were performed. The tests follow current peer-reviewed published methods for assessing the effects of biologically active compounds on human neuronal cells. The in vitro study showed a significant improvement in cell viability and reactive oxygen species (ROS) inhibition using the Braini® compounds.

Based on existing published science supporting the neuroprotective role of the Braini® formulation, this supplement may be useful and to improve cognitive function and health. Based on studies conducted outside the United States, the research team hypothesizes that orally ingested Braini® taken as directed (2 x 525 mg powdered capsules per day), will demonstrate superior improvements in standardized cognitive performance assays. MOCA scores will be used for screening patients. The research team aims to conduct a randomized, placebo-controlled, double-blinded dietary supplement study to evaluate this hypothesis among a cohort of younger and a cohort of older healthy adults.

ELIGIBILITY:
Inclusion Criteria:

1. 18-30 or 55-80 years of age
2. Agree to continue with current diet and refrain from taking any new nutritional or herbal supplements
3. Willing to participate in the trial for 30-35 days, including taking a placebo
4. Able to understand and write English

Exclusion Criteria:

1. Clinically diagnosed with Alzheimer's disease, stroke, Parkinson's disease, or dementia
2. Taking prescription drugs to support memory/prevent cognitive decline in the past 180 days or to treat other diseases referenced below in criterion number.
3. Taking dietary supplements that include wild blueberry extract, Neurxcel, or silk portein peptide in the past 90 days
4. Active fibromyalgia, multiple sclerosis, seizures/epilepsy or other known diseases that affect memory or cognition
5. Taking an medicines that are stimulants including Adderall XR (amphetamine), Concerta (methylphenidate), Dexedrine (amphetamine), Evekeo (amphetamine), Focalin XR (methylphenidate), Quillivant XR (methylphenidate), Ritalin (methylphenidate), Strattera (atomoxetine hydrochloride), or Vyvanse (lisdexamfetamine dimesylate).
6. GI disorders known to impair absorption of nutrients
7. Traumatic brain injury (TBI) in personal history
8. MOCA test score <21
9. Pregnancy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2020-04-09 (Actual); Study Completion 2020-04-30 (Actual)

PRIMARY OUTCOMES:
CNS Vital Signs test battery | 28 days
  The CNS Vital Signs test is a computerized neuropsychological battery that includes seven sub-tests designed to screen cognitive abilities. The Verbal Memory Test involves immediate and delayed recognition for words presented on the screen. The Visual Memory Test involves immediate and delayed recognition of geometric figures. The Finger Tapping Test involves rapidly press the space bar. The Symbol Digit Coding Test involves typing numbers that correspond to different symbols presented on screen. The Stroop Test contains three parts that involve responding to words and colors. The Shifting Attention Test involves matching geometric objects either by shape or by color. The Continuous Performance Test is a 5-min sustained attention test that involves responding to the target stimulus. Results are given as normed domain scores for Memory, Psychomotor Speed, Reaction Time, Complex Attention, and Cognitive Flexibility each with a mean score of 100 and SD of 15

CONTACTS AND LOCATIONS:
Overall Officials: Amy J Lanou, PhD, Principal Investigator — UNC Asheville
Locations (1):
- University of North Carolina at Asheville, Asheville, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No
Upon starting the study, participants will be given an ID number, and the informed consent document will be separated from their file. Only study personnel will have access to both names and ID numbers. Data will be entered into a data management file (Excel and then SPSS) that will be kept on a password-protected computer. Data will be kept for three years and then destroyed (deleted and shredded).

REFERENCES:
- [Derived] Lanou AJ, Mast AC, Hill BD, Kim SS, Hanaway P. A Randomized, Placebo-Controlled Clinical Trial of a Novel Dietary Supplement on Standardized CNS Vital Signs Cognitive Performance Parameters in Adults. J Integr Complement Med. 2023 May;29(5):303-312. doi: 10.1089/jicm.2022.0543. Epub 2023 Feb 28. PMID 36856456